CLINICAL TRIAL: NCT00004464
Title: High Dose Cyclophosphamide for the Treatment of Severe Aplastic Anemia and Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Study of High Dose Cyclophosphamide in Patients With Severe Aplastic Anemia and Paroxysmal Nocturnal Hemoglobinuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: J9611; 96-01-17-02 (Other: JHM IRB); JHOC-96011702; JHOC-9611 (Other: other); 199/13895 (Other: other)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2018-08

CONDITIONS: Aplastic Anemia; Paroxysmal Hemoglobinuria, Nocturnal
Keywords: aplastic anemia; hematologic disorders; paroxysmal nocturnal hemoglobinuria; rare disease
MeSH Terms: conditions — Anemia, Aplastic; Hemoglobinuria, Paroxysmal; Hematologic Diseases; Rare Diseases | interventions — Cyclophosphamide; Filgrastim

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: cyclophosphamide
Drug: filgrastim

SUMMARY:
OBJECTIVES: I. Confirm the efficacy demonstrated in a pilot study using high dose cyclophosphamide in patients with severe aplastic anemia.

II. Determine whether the addition of filgrastim (G-CSF) to high dose cyclophosphamide shortens the time to recovery in these patients.

III. Determine whether this regimen is efficacious in treating paroxysmal nocturnal hemoglobinuria.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive high dose cyclophosphamide IV on days 1-4. Beginning on day 10, patients receive filgrastim (G-CSF) until the absolute neutrophil count is greater than 1,000/mm3 for 2 consecutive days.

Patients are followed every 3 months for at least 2 years and annually thereafter.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Acquired severe aplastic anemia or paroxysmal nocturnal hemoglobinuria
* Not a candidate for allogeneic bone marrow transplantation
* Must meet one of the following criteria:

  * Severe aplastic anemia

    * Less than 25% bone marrow cellularity and depression in two of three blood counts (reticulocytes less than 40,000/mm3
    * platelet count less than 20,000/mm3 and granulocytes less than 500/mm3)
  * Life-threatening paroxysmal nocturnal hemoglobinuria

    * Absolute neutrophil count less than 500/mm3
    * platelet transfusion dependent
    * thrombotic disease
* No Fanconi anemia
* No abnormal cytogenetics

--Patient Characteristics--

* Renal: Creatinine no greater than 2.0 mg/dL
* Cardiovascular: Cardiac ejection fraction at least 45%
* Other: Not preterminal or moribund Not pregnant

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 1996-02; Primary Completion 2007-03-01 (Actual); Study Completion 2008-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Brodsky, Study Chair — Johns Hopkins University
Locations (1):
- Johns Hopkins Oncology Center, Baltimore, Maryland, United States